CLINICAL TRIAL: NCT04057794
Title: Parkinson's Foundation: PD Generation: Mapping the Future of Parkinson's Disease
Brief Title: PDGeneration: Mapping the Future of Parkinson's Disease
Acronym: PDGENE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Parkinson's Foundation (Other)
Collaborators: Fulgent Laboratories (Unknown); Indiana University (Other); The Parkinson Study Group (Network); Navitas Clinical Research, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: PDGene-01
Record Dates: First submitted 2019-08-06; First posted 2019-08-15 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Parkinson's Disease and Parkinsonism
Keywords: Parkinson's; Genetics; PD Genetics
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: All participants will undergo genetic counseling service post-genetic testing either locally or through central services.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Site-Based Genetic Counseling (Active Comparator): Participants randomized to this arm will receive genetic counseling for genetic results through the enrolling site.
  Interventions: Device: Lab Assay for seven genetic variants for Parkinson's Disease
- Centralized Genetic Counseling (Active Comparator): Participants randomized to this arm will receive genetic counseling for genetic results through a centralized genetic counseling group at Indiana University.
  Interventions: Device: Lab Assay for seven genetic variants for Parkinson's Disease

INTERVENTIONS:
Device: Lab Assay for seven genetic variants for Parkinson's Disease — Counseling provided to participant by site clinician/physician/genetic counselor.
  Arms: Site-Based Genetic Counseling
Device: Lab Assay for seven genetic variants for Parkinson's Disease — Counseling provided to participant by centralized genetic counseling group at Indiana University.
  Arms: Centralized Genetic Counseling

SUMMARY:
To assess the feasibility, impact, and participant satisfaction of offering Clinical Laboratory Improvement Amendments (CLIA) certified genetic testing as part of clinical care for People with Parkinson's disease (PWP).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate how offering Clinical Laboratory Improvement Amendments (CLIA) certified genetic testing for Parkinson's Disease (PD) genes to people with Parkinson's Disease impacts clinical care and potential enrollment in clinical trials. This multi-center study will assess the impact and satisfaction of the mode of genetic counseling by comparing counseling conducted by a clinician versus centralized genetic counseling conducted through Indiana University. The study will also assess knowledge gained by administering a knowledge survey pre- and post-genetic testing. All genetic test results will be returned to participants through a genetic counseling visit.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's Disease: probable diagnosis.
2. Willingness to undergo genetic testing, and choose to be informed of genetic testing results for Glucosylceramidase Beta (GBA), LRRK2 and 5 additional PD related genes (SNCA, VPS35, PRKN, PINK-1, PARK7).
3. Capacity to give full informed consent in writing, and have read and signed the informed consent forms (ICFs) based on clinician's determination.
4. Able to perform study activities (including completion of either online, in-person or paper surveys).
5. Individuals must speak and understand the language of the informed consent.

Exclusion Criteria:

1. Diagnosis of an atypical parkinsonian disorder (i.e., multiple system atrophy, progressive supranuclear palsy, dementia with Lewy bodies, corticobasal syndrome), including that due to medications, metabolic disorders, encephalitis, cerebrovascular disease, or normal pressure hydrocephalus.
2. Individuals who have received a blood transfusion within the past 3 months.
3. Individuals who have active hematologic malignancies such as lymphoma or leukemia.
4. Individuals who have had a bone marrow transplant within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1982 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of genetic testing and counseling | up to 24 weeks
  The total number of participants who receive genetic testing and counseling.
Impact Evaluation | up to 6 months
  The impact of knowledge gained by people with Parkinson's by assessing returned survey responses regarding their behavior and follow-up to clinical care after receipt of genetic counseling.
Satisfaction Comparison | up to 6 months
  Differences in satisfaction of receiving genetic test results and genetic counseling by enrolling site (clinician/genetic counselor) or centralized counseling group using the Clinical Genetic Counseling Satisfaction Score.

SECONDARY OUTCOMES:
Number of participants that enroll in precision medicine trials | up to 12 months
  Number of participants that enroll in precision medicine trials
Time it takes between first contact to the return of genetic test results | up to 12 months
  Number of weeks it takes between participant consent to return of genetic test results.

CONTACTS AND LOCATIONS:
Overall Officials: Roy N Alcalay, MD, MS, Principal Investigator — Columbia University
Locations (13):
- United States (13):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of California San Diego (UCSD), La Jolla, California
  - University of Miami, Fort Lauderdale, Florida
  - Cleveland Clinic Florida-Weston, Weston, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Health Partners/Park Nicollet: Struthers Parkinson's Center, Minneapolis, Minnesota
  - Beth Israel Medical Center, New York, New York
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- See also: For more information and to enroll, please visit the website. — http://www.parkinson.org/PDGENEration

DOCUMENTS (1):
  • Informed Consent Form (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT04057794/ICF_000.pdf